CLINICAL TRIAL: NCT01316731
Title: Effects of Acute Exercise on (Myokine) Gene Expression in Human Skeletal Muscle
Brief Title: MyoGene: Effects of Acute Exercise on (Myokine) Gene Expression in Human Skeletal Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Dutch Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL33968.081.10
Record Dates: First submitted 2011-03-10; First posted 2011-03-16 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Exercise; Muscle; Gene Expression; Myokine
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental)
  Interventions: Other: Single legged exercise

INTERVENTIONS:
Other: Single legged exercise — A single exercise bout that consists of one hour one-legged cycling on a adapted recumbent cycle ergometer at a submaximal rate. The non-exercising leg will serve as control for the exercising leg.

SUMMARY:
Rationale: Proteins released from muscle during and shortly after exercise, often referred to as myokines, may be central to our understanding of the cross-talk during and after exercise between skeletal muscles and other organs, in particular the liver. So far only a few myokines are identified (e.g. IL-6, IL-8, IL-15, TNF-alpha). Taking into account the role of these several known myokines in developing insulin resistance, revealing new putative myokines might provide valuable information and a direction for future research on the pathogenesis and treatment of type 2 diabetes mellitus.

Objective: The objective of the present study is to identify novel myokines, expression of which is altered in skeletal muscle after a single bout of exercise.

Study design: experimental study. Study population: Ten healthy, male subjects between 40 and 60 years of age and BMI < 30 kg/m2, will participate in this study.

Intervention: A single exercise bout that consists of one hour one-legged cycling on a adapted recumbent cycle ergometer at a submaximal rate. The non-exercising leg will serve as control for the exercising leg.

Main study outcomes: Main study outcomes include upregulation of genes in skeletal muscle after exercise (with a focus on genes encoding myokines) and changes of blood plasma levels of selected proteins after exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-60 years
* Male gender
* BMI < 30 kg/m2

Exclusion Criteria:

* Exercising regularly (> 2 times a week, > 3 hour in total per week)
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Following, or have recently followed a (weight-loss) diet
* Donated or intended to donate blood 2 months before until two months after the study
* Medical condition that can interfere with the study outcome (i.e. cardiovascular disease, pulmonary disease)
* Systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg
* Use of medications known to interfere with gene expression in the muscles (i.e. statins, fenofibrate).
* Use of antithrombotic therapy (marcoumar, sintromitis).
* Diagnosed diabetes mellitus type 1 or 2.
* Drugs or alcohol abuse ( > 3 glasses of alcoholic beverages a day).
* (Chronic) injuries of the locomotor system that can interfere with the intervention
* Participated in another study within the last six months

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Gene expression changes in skeletal muscle from baseline to after exercise | T = 0 and T =1
  Gene expression is measured using whole genome Affymatrix microarrays Muscle tissue will be collected at time points T = 0 (before exercise) and T = 1 (directly after exercise). Special focus is on the changes in genes coding for myokines. Up to 5 genes will be selected for follow-up analysis.
Changes in plasma levels of selected proteins | T = 0, T =1 and T = 3
  Selected proteins will be analyzed by ELISA assays or western blot analysis, depending on ELISA availability at T = 0, T = 1 and T = 3 (2 hours post-exercise). The selection of the proteins is based on significance, the robustness of induction (>80% of subjects showing induction) and the magnitude of the induction ( mean fold change > 2)

SECONDARY OUTCOMES:
PBMC gene expression changes before and after exercise | T = 0, T = 1 and T =3
  Gene expression changes in the blood will be assessed using whole genome Affymetrix microarrays for the samples at T = 0, 1 and 3.
Routine plasma level changes before and after exercise | T = 0, 1 and 3
  At all three time point (T = 0, 1 and 3) plasma levels of glucose, insulin, fatty acids, triglycerides, cortisol, adrenalin and lactate will be determined.
Heart rate changes, baseline compared with exercise | During the intervention
  Heart rate will be measured during the maximum work load test and the experimental exercise period.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Human Nutrition, Wageningen University, Wageningen, Gelderland, Netherlands